CLINICAL TRIAL: NCT00376519
Title: Umbilical Cord Blood Transplant With Co-Infusion of T Regulatory Cells
Brief Title: Umbilical Cord Blood T-Regulatory Cell Infusion Followed by Donor Umbilical Cord Blood Transplant in Treating Patients With High-Risk Leukemia or Other Hematologic Diseases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMN-2005LS011; UMN-0502M67473 (Other: IRB, University of Minnesota); UMN-MT2005-01 (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Secondary Myelofibrosis
Keywords: graft versus host disease; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; secondary acute myeloid leukemia; refractory anemia with excess blasts; myelodysplastic syndromes; chronic myelogenous leukemia; refractory anemia; prolymphocytic leukemia; stage IV adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; follicular lymphoma; mantle cell lymphoma; chronic idiopathic myelofibrosis; secondary myelofibrosis; refractory chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma; recurrent marginal zone lymphoma; marginal zone lymphoma; diffuse large cell lymphoma; anaplastic large cell lymphoma; lymphoblastic lymphoma; immunoblastic large cell lymphoma; multiple myeloma
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Refractory; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Primary Myelofibrosis; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large-Cell, Immunoblastic | interventions — Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant with Treg Cells (Experimental): Patients receive preparative therapy with Fludarabine, cyclophosphamide, total body irradiation and Treg infusion followed by umbilical cord blood transplantation.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Procedure: Treg cell infusion; Procedure: umbilical cord blood transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Drug: cyclophosphamide — Cyclophosphamide 60 mg/kg/day will be administered as a 2 hour intravenous infusion with a high volume fluid flush and mesna (MT(S)9006) on day -8 and -7 one hour after fludarabine infusion.
  Other Names: Cytoxan
Drug: cyclosporine — Will be administered beginning on day -3 and adjusted to maintain a level of >200. For adults the initial dose will be 2.5 mg/kg intravenously (IV) over 2 hours every 12 hours.
  Other Names: CSA
Drug: fludarabine phosphate — Fludarabine 25 mg/m^2/day will be administered as a 1 hour intravenous infusion on days -9 through -7.
  Other Names: Fludara
Drug: mycophenolate mofetil — All patients will begin mycophenolate mofetil (MMF) on day -3, at the dose of 3 grams/day divided into 2 or 3 doses (every 12 or 8 hours).
  Other Names: MMF
Procedure: Treg cell infusion — On day -1 prior to UCB transplantation, Treg cells will be infused IV without in-line filtration. A semi-log dose escalation of CD4+CD25+ Treg cells is scheduled with 3 patients at each step. Doses will be 0.1 x 10^6/kg, 0.3 x 10^6/kg, 1 x 10^6/kg and 3 x 10^6/kg weight (determined on the day prior to administration of the preparative therapy).
Procedure: umbilical cord blood transplantation — Following the administration of the preparative therapy, all subjects will undergo UCB transplantation. The UCB will be administrated by IV infusion without in-line filtration.
  Other Names: UCBT
Radiation: total-body irradiation — Radiotherapy: 165 cGy will be administered on day -5 through -2 two fractions each day.

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine and cyclophosphamide, and total-body irradiation before a donor umbilical cord blood stem cell transplant helps stop the growth of cancer or abnormal cells and prepares the patient's bone marrow for the stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer or abnormal cells (graft-versus-tumor effect). Giving an infusion of the donor's T-regulatory cells before the transplant may help increase this effect. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of umbilical cord blood T-regulatory cell infusion followed by donor umbilical cord blood transplant in treating patients with high-risk leukemia or other hematologic diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of umbilical cord blood (UCB)-derived CD4- and CD25-positive T-regulatory (Treg) cell infusion followed by double unrelated donor UCB transplantation in patients with high-risk leukemia or other hematologic diseases.

Secondary

* Determine the speed of neutrophil and platelet recovery at day 42 in these patients.
* Determine the incidence of "double chimerism" (e.g., engraftment of both UCB units) at day 21 in these patients.
* Determine the risk of severe grade III-IV acute graft-versus-host disease (GVHD) at day 100 in these patients.
* Determine the risk of chronic GVHD at 1 year post transplantation in these patients.
* Determine the probability of survival at 100 days and 1 year post transplantation in these patients.

OUTLINE: This is an open-label, dose-escalation study of CD4- and CD25-positive umbilical cord blood (UCB)-derived T-regulatory cells (Treg).

* Preparative therapy: Patients receive fludarabine phosphate intravenously (IV) over 1 hour on days -9 to -7 and cyclophosphamide IV over 2 hours on days -8 and -7 (1 hour after fludarabine infusion). Patients then undergo total-body irradiation (TBI) twice daily on days -5 to -2.
* UCB-derived Treg infusion: Patients receive UCB-derived Treg cells IV on day -1.
* Double unrelated donor UCB transplantation: Patients undergo double unrelated donor UCB transplantation by IV infusion on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV over 2 hours or orally 2 or 3 times daily beginning on day -3 and continuing until day 100, followed by a taper to day 180, in the absence of GVHD. Patients also receive mycophenolate mofetil (MMF) orally or IV twice daily on days -3 to 30 or 7 days after engraftment, whichever is later, in the absence of acute GVHD*. If no donor engraftment occurs, MMF may be continued at the discretion of the attending physician.

NOTE: *If the patient has acute GVHD requiring systemic therapy, MMF may be stopped 7 days after GVHD is controlled (e.g., resolution of skin rash, vomiting, and diarrhea).

Cohorts of 3-6 patients receive escalating doses of UCB-derived Treg cells until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience nonhematologic dose-limiting toxicity within 48 hours of Treg cell infusion. At least 6 patients are treated at the MTD.

ELIGIBILITY:
Inclusion Criteria:

Patient and Donor Demographic Criteria

* Patient must be 18-45 years of age.
* Patients must have three partially HLA matched UCB units. Units identified as the HSC source must be HLA matched at 4-6 HLA- A and B (at low to intermediate resolution) and DRB1 (at high resolution), and the units must be HLA matched at 4-6 HLA- A, B, DRB1 antigens with each other. Total cryopreserved HSC graft cell dose must be >2.5 x 107 nucleated cells per kilogram recipient body weight. Also, the two umbilical cord blood (UCB) units must be ABO-matched.
* The UCB unit identified as the Treg source must be HLA matched at 4-6 HLA antigens with the patient (without an HLA or ABO matching criterion with the UCB HSC source).

Disease Criteria

* Patients must have a hematological malignancy as listed below:

  * Acute myelogenous leukemia: high risk CR1 (as evidenced by preceding myelodysplastic syndrome (MDS), high risk cytogenetics such as those associated with MDS or complex karyotype, or >2 cycles to obtain complete remission (CR); second or greater CR. Must be in remission by morphology (<5% blasts within normocellular marrow).
* Acute lymphocytic leukemia: high risk CR1 as evidenced by high risk cytogenetics [t(9;22), t (1:19), t(4;11) or other MLL rearrangements] or > 1 cycle to obtain CR; second or greater CR.
* Chronic myelogenous leukemia resistant to imatinib therapy
* Myelodysplasia (MDS) IPSS Int-2 or High risk (i.e. RAEB, RAEBt) or refractory anemia with severe pancytopenia or high risk cytogenetics. Blasts must be < 10% by a representative bone marrow aspirate morphology (otherwise induction chemotherapy to achieve < 10% blasts is required pre-transplant).
* Advanced myelofibrosis
* Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma or follicular lymphoma that have progressed after at least two prior therapies. Patients with bulky disease (nodal mass greater than 5 cm) should be considered for debulking chemotherapy before transplant.
* Lymphoplasmacytic lymphoma, mantle-cell lymphoma, prolymphocytic leukemia are eligible after initial therapy in CR1+ or PR1+.
* Large cell non-Hodgkins lymphoma (NHL) > CR2/> PR2. Patients in CR2/PR2 with initial short remission(<6 months) are eligible.
* Lymphoblastic lymphoma, Burkitt's lymphoma, and other high-grade NHL after initial therapy if stage III/IV in CR1/PR1 or after progression if stage I/II <1 year.
* Multiple myeloma beyond PR2. Patients with chromosome 13 abnormalities, first response lasting less than 6 months, or β-2 microglobulin > 3 mg/L, may be considered for this protocol after initial therapy.
* Recipients will have a Karnofsky score > 80% and have acceptable organ function ie creatinine < 2.0, bilirubin, AST/ALT, ALP < 2 x normal, pulmonary function > 50% normal, left ventricular ejection fraction > 45%. Note: All patients with a creatinine > 1.2 or a history of renal dysfunction must have creatinine clearance (must be > 40 ml/min to be eligible).
* Recipients will sign informed consent approved by the Committee on the Use of Human Subjects at the University of Minnesota.

Exclusion Criteria:

* Pregnant or breastfeeding
* Evidence of HIV infection or known HIV positive serology
* Current active infection
* Available HLA matched sibling donor.
* CML in active blast crisis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of T-regulatory cells | Within 24 Hours
  Dose limiting toxicities (DLT) are defined as any grade 3-4 toxicity within 24 hours of Treg cell infusion, excluding hematological .

SECONDARY OUTCOMES:
Incidence of neutrophil recovery | Day 42
Incidence of double chimerism | Day 21
Incidence of grades II-IV and III-IV acute graft-versus-host disease (GVHD) | Day 100
Incidence of chronic graft-versus-host disease | 1 Year
Survival | Day 100 and 1 Year
Incidence of Platelet Recovery | Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G. Brunstein, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States